CLINICAL TRIAL: NCT06688058
Title: A Phase 1, Randomized, Double-Blind, Comparator-Controlled, Dose-Escalation Trial to Evaluate, Tolerability, and Immunogenicity of V540D in Healthy Adults.
Brief Title: A Trial to Evaluate Tolerability and Immunogenicity of V540D in Healthy Adults (V540D-004)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: V540D-004
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Healthy
MeSH Terms: interventions — Neu1 protein, mouse

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- V540D (Experimental): Participants will receive vaccinations with V540D.
  Interventions: Biological: V540D
- GARDASIL®9 (Active Comparator): Participants will receive vaccinations with GARDASIL®9.
  Interventions: Biological: GARDASIL®9

INTERVENTIONS:
Biological: V540D — Experimental vaccine and adjuvant administered via intramuscular (IM) injection
  Arms: V540D
Biological: GARDASIL®9 — Suspension administered via IM injection
  Other Names: G9; V503
  Arms: GARDASIL®9

SUMMARY:
Researchers are looking for new ways to prevent cancers related to human papillomavirus (HPV). HPV is a common virus that can cause an infection. There are many different types of HPV. Most people's immune system can fight HPV infection and it goes away without treatment. For some people, HPV infections can last longer and may cause cancer years later.

A standard vaccine to prevent HPV-related cancers is GARDASIL®9 (G9). G9 protects against 9 types of HPV but it does not protect against other types of HPV. The study vaccine (called V540D) is designed to protect against the same HPV types that G9 protects against plus other HPV types. The main goal of this study is to learn about the safety of V540D in healthy adults and if people tolerate it.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Is in good health based on medical history, physical examination, vital sign (VS) measurements and electrocardiograms (ECGs) performed before randomization

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a history of abnormal Pap smears, HPV- related external genital lesions (eg, condyloma acuminate, vulval intraepithelial neoplasia (VIN), or prostatic intraepithelial neoplasia (PIN)) or external genital cancer (eg, penile cancer), HPV-related vaginal or anal lesions (eg, condyloma acuminata or vaginal intraepithelial neoplasia (VaIN)) or vaginal or anal cancer
* Has a history of cancer (malignancy)
* Has received any HPV vaccine or is expected to receive any HPV vaccine during the study, outside the protocol

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience a Solicited Injection-Site Adverse Event (AE) | Up to approximately 6 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants Who Experience a Solicited Systemic AE | Up to approximately 6 months
  Solicited systemic AEs include headache, fatigue, nausea, dizziness, muscle aches, joint pain.
Number of Participants Who Experience Immediate Reactions Occurring Within 30 Minutes After Any Vaccination | Up to approximately 6 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants Who Experience Unsolicited AEs | Up to approximately 7 months
  An unsolicited AE is an event that is not predefined as a solicited AE or is predefined as a solicited AE but reported at any time outside the solicited time period.
Number of Participants Who Experience a Serious Adverse Event (SAE) | Up to approximately 18 months
  SAEs include AEs that result in any of the following outcomes: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect.
Number of Participants Who Experience a Medically-Attended AE (MAAE) | Up to approximately 18 months
  AEs in which medical attention is received during an unscheduled, non-routine outpatient visit, such as an emergency department visit, office visit, or an urgent care visit with any medical personnel for any reason. Routine visits are not considered MAAEs. Examples of routine visits include physical examination, wellness visits, or vaccinations.
Number of Participants Who Experience an Event of Clinical Interest (ECI) | Up to approximately 18 months
  ECIs are defined as an overdose of Sponsor's product, drug-induced liver injury events, or potential immune-mediated diseases (pIMDs).

SECONDARY OUTCOMES:
Total Immunoglobulin G (IgG) Geometric Mean Ratios (GMRs) for anti-HPV types 6, 11, 16, 18, 31, 33, 45, 52, and 58 | Up to approximately 7 months
  GMR of titers for participants vaccinated with V540D versus those who received GARDASIL®9 alone will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (4):
- United States (4):
  - Research Centers of America ( Hollywood ) ( Site 0001), Hollywood, Florida
  - Velocity Clinical Research, Savannah ( Site 0005), Savannah, Georgia
  - Alliance for Multispecialty Research, LLC ( Site 0003), Kansas City, Missouri
  - Alliance for Multispecialty Research, LLC ( Site 0004), Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com